CLINICAL TRIAL: NCT04870502
Title: Effect of Ubiquinol Supplementation on Ovulation Induction in Clomiphene Citrate Resistance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saudi German Hospital - Madinah (Other)
Responsible Party: Principal Investigator, Islam Mohamed Magdi Ammar, Associate Professor and Consultant of Obstetrics and Gynecology, Saudi German Hospital - Madinah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGHM-MAR2019-OBGYN
Record Dates: First submitted 2021-04-09; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clomiphene citrate and Ubiquinol (Active Comparator): Controlled ovarian stimulation (COS) was done by Clomiphene Citrate (Fertab® 50 mg tablets, Zynova. SITCO Pharma.) as 150 mg (3 tablets) daily for 5 days (from 2nd day till 6th day of the cycle) together with Ubiquinol (active form of Coenzyme Q10) starting from 2nd day till the day of human Chorionic Gonadotropin (hCG) triggering in a dose of 100 mg capsules orally once daily, immediately after meal (Nutraquinol®; Jamjoom Pharma Nutraceuticals).
  Interventions: Drug: Controlled ovarian stimulation by Combined Clomiphene Citrate and Ubiquinol Versus hMG
- Human Menopausal Gonadotropins (hMG) (Active Comparator): Controlled ovarian stimulation (COS) was done by Human Menopausal Gonadotropins (hMG) (Merional® 75 I.U. vials, IBSA.) IM was given from 2nd day of the cycle in a dose ranging from 75 to 225 IU according to the patient's response.
  Interventions: Drug: Controlled ovarian stimulation by Combined Clomiphene Citrate and Ubiquinol Versus hMG

INTERVENTIONS:
Drug: Controlled ovarian stimulation by Combined Clomiphene Citrate and Ubiquinol Versus hMG — In group A, controlled ovarian stimulation (COS) was done by Clomiphene Citrate (Fertab® 50 mg tablets, Zynova. SITCO Pharma.) as 150 mg (3 tablets) daily for 5 days (from 2nd day till 6th day of the cycle) together with Ubiquinol (active form of Coenzyme Q10) starting from 2nd day till the day of human Chorionic Gonadotropin (hCG) triggering in a dose of 100 mg capsules orally once daily, immediately after meal (Nutraquinol®; Jamjoom Pharma Nutraceuticals). In group B, Human Menopausal Gonadotropins (hMG) (Merional® 75 I.U. vials, IBSA.) IM was given from 2nd day of the cycle in a dose ranging from 75 to 225 IU according to the patient's response. Patients were instructed not to take any non-study drugs during the whole study period.
  Other Names: Fertab® 50 mg tablets, Zynova. SITCO Pharma.; Nutraquinol®; Jamjoom Pharma Nutraceuticals; Merional® 75 I.U. vials, IBSA

SUMMARY:
Objective: To evaluate potential benefits of adding the active form of Coenzyme Q10 (Ubiquinol) to Clomiphene Citrate compared with Human Menopausal Gonadotropins (hMG) in Clomiphene Citrate resistant PCOS patients.

Methods: 148 PCOS Patients with Clomiphene Citrate resistance were randomized into two groups (A and B). In group A, controlled ovarian stimulation was done by Clomiphene Citrate 150 mg daily (from 2nd till 6th day of cycle) together with Ubiquinol starting from 2nd day till day of hCG triggering in a dose of 100 mg orally once daily. In group B, hMG was given from 2nd day of the cycle in a dose ranging from 75 to 225 IU. Serial transvaginal ultrasonography was done starting on cycle day 8 and continued till size of leading follicle reaches 18 mm or more then ovulation triggering was done. Thereafter, patients were advised for a timed intercourse (TI) after 36 hours. A blood sample was withdrawn seven days after hCG triggering, for measurement of serum progesterone. If the Patient presented with a missed period for one week, a serum sample was sent for β-hCG.

DETAILED DESCRIPTION:
Patients were divided randomly into two groups (A and B), who underwent controlled ovarian stimulation and timed intercourse, using random table computer software (Open Epi version 3.21).

Basal transvaginal ultrasonography (TVS) was done on day 2 of the cycle before commencing ovarian stimulation. For patients presenting with amenorrhea or oligomenorrhea, dydrogesterone 10 mg (Duphaston®; Abbott Biologicals B.V.) was prescribed (3 times daily for 10 days) to achieve withdrawal bleeding before starting induction of ovulation.

In group A, controlled ovarian stimulation (COS) was done by Clomiphene Citrate (Fertab® 50 mg tablets, Zynova. SITCO Pharma.) as 150 mg (3 tablets) daily for 5 days (from 2nd day till 6th day of the cycle) together with Ubiquinol (active form of Coenzyme Q10) starting from 2nd day till the day of human Chorionic Gonadotropin (hCG) triggering in a dose of 100 mg capsules orally once daily, immediately after meal (Nutraquinol®; Jamjoom Pharma Nutraceuticals). In group B, Human Menopausal Gonadotropins (hMG) (Merional® 75 I.U. vials, IBSA.) IM was given from 2nd day of the cycle in a dose ranging from 75 to 225 IU according to the patient's response. Patients were instructed not to take any non-study drugs during the whole study period. All patients did not receive any drug for induction of ovulation 3 months prior to participation in the study.

Serial transvaginal ultrasonography was done for assessment of follicular growth (number and diameter of follicles) and endometrial thickness (measured on sagittal view of the uterus by including the whole endometrium at the point of its maximum thickness), starting on cycle day 8, using vaginal 4.5 MHz endocavity transducer (Esaote Mylab 50 Xvision Ultrasound, Italy), and was continued with an interval of 1-3 days till the size of the leading follicle reaches 18 mm or more in mean follicular diameter. Then ovulation triggering was done by an intramuscular single dose of human Chorionic Gonadotropin (Epifasi® 5000 IU vials, EIPICO, Egypt.) 2 vials (10,000 IU). Thereafter, patients were advised for a timed intercourse (TI) 36 hours after ovulation triggering.

All measurements were obtained by a blinded single operator. All data were digitally stored and were not analyzed till the end of the study.

Thereafter, patients were asked to come for follow up, 7 days after hCG triggering, where a blood sample (2 mL) was withdrawn for measurement of serum progesterone (ng/ml). Collected samples were centrifuged and then stored at 2-8 °C until enzyme immunoassay was done. If the Patient presented with a missed period for a week, a serum sample was sent for β-hCG using immunoassay.

Patients with positive serum pregnancy test, defined as β-hCG concentration >10 mU/ml, were examined by abdominal ultrasonography 6 weeks after the first day of their last menstrual period with 3.5 MHz sector transducer (Esaote Mylab 50 Xvision Ultrasound, Italy) to detect an intrauterine gestational sac (Clinical pregnancy). Patients who failed to get pregnant were requested for follow up for 2 more consecutive cycles with the same protocol.

The primary outcomes measured were; number of cases achieving follicular growth to the size of mature follicle ≥ 18 mm (1-3 follicles) during the three cycles of stimulation, number of stimulated cycles (till pregnancy occurs or completing the 3 cycles of the study, whichever is earlier), the endometrial thickness on the day of triggering, and the luteal function as assessed by mid-luteal serum progesterone measurements.

The secondary outcomes were; number of cases with positive serum pregnancy test and the clinical pregnancy rate among the two groups during the three cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with Clomiphene Citrate resistant PCOS who fulfilled the following inclusion criteria:

* Age 18 to 35 years
* Body mass index (BMI) between 18.5 and 34.9 kg/m2
* Presenting with primary or secondary infertility.

PCOS was diagnosed according to the Rotterdam ESHRE/ASRM Consensus workshop, with at least 2 of the following 3 criteria:

A- Oligo- and/or anovulation; manifested by oligomenorrhea or amenorrhea. Oligomenorrhea was defined as cycle interval of more than 35 days but less than six months. Amenorrhea was defined as absence of menstruation for six months or more.

B- Hyperandrogenism; biochemical and/or clinical in the form of acne or hirsutism defined as a score of 8 or higher using the modified Ferriman-Gallwey scoring system when abnormal hair distribution was assessed in nine body areas and given a score of 0 to 4.

C - Polycystic ovarian morphology detected by transvaginal ultrasound with the presence of 12 or more follicles measuring 2-9 mm in diameter in one or both ovaries, and/or increased ovarian volume >10 mL.

* Clomiphene Citrate resistance was defined as failure of ovulation after administration of Clomiphene Citrate in a dose of 150 mg for 5 days per cycle, for two or three cycles.
* Patent both fallopian tubes and normal uterine cavity as evidenced by hysterosalpingography (HSG).
* Their partners had normal semen parameters as defined by the modified WHO 2010 criteria.

Exclusion criteria were:

* Morbidly obese patients with BMI ≥35 Kg/2m.
* Abnormal husband semen analysis.
* Abnormal HSG or laparoscopic evidence of pelvic adhesions.
* Patients receiving statin drugs for cholesterol, beta-blockers for high blood pressure, or tricyclic antidepressants, were also excluded as these drugs can lower the levels of ubiquinol in the body.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change of the number of cases achieving follicular growth to the size of mature follicle ≥ 18 mm (1-3 follicles) during the three cycles of stimulation | The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
  Serial transvaginal ultrasonography was done for assessment of follicular growth (number and diameter of follicles) starting on 8th day of the menstrual cycle, using vaginal 4.5 MHz endocavity transducer (Esaote Mylab 50 Xvision Ultrasound, Italy), and is continued with an interval of 1-3 days till the size of the leading follicle reaches 18 mm or more in the mean follicular diameter. The mean follicular diameter (MFD) is calculated by summation of the length and width of the growing follicle, divided by two. Mature follicle is defined as a follicle with mean diameter of 18-22 mm. The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
Change of the number of stimulated cycles (till pregnancy occurs or completing the 3 cycles of the study, whichever is earlier). | The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
  Controlled ovarian stimulation is carried out for 3 menstrual cycles. Each menstrual cycle is of 3-5 weeks duration. The estimated period of time is 3 menstrual cycles (total of 9-15 weeks) or till pregnancy occurs whichever came first.
Change of Luteal function as assessed by mid-luteal serum progesterone measurements. | The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
  Patients were asked to come for follow up, 7 days after hCG triggering, where a blood sample (2 mL) was withdrawn for measurement of serum progesterone (ng/mL). Collected samples were centrifuged and then stored at 2-8 °C until enzyme immunoassay was done. Normal luteal function was defined as mid-luteal serum progesterone levels > 10 ng/mL. This is carried out for 3 menstrual cycles of controlled ovarian stimulation. Each menstrual cycle is of 3-5 weeks duration. The estimated period of time is 3 menstrual cycles (total of 9-15 weeks) or till pregnancy occurs whichever came first.
Change of Endometrial thickness (mm) on the day of hCG triggering | The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
  Transvaginal ultrasonography was done for assessment of endometrial thickness in mm (measured on sagittal view of the uterus by including the whole endometrium at the point of its maximum thickness) on the day of hCG triggering using vaginal 4.5 MHz endocavity transducer (Esaote Mylab 50 Xvision Ultrasound, Italy). This is carried out for 3 menstrual cycles of controlled ovarian stimulation. Each menstrual cycle is of 3-5 weeks duration. The estimated period of time is 3 menstrual cycles (total of 9-15 weeks) or till pregnancy occurs whichever came first.

SECONDARY OUTCOMES:
Change of the number of cases with positive serum pregnancy test (Chemical pregnancy) | The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
  If the Patient presented with a missed period for a week, a serum sample was sent for β-hCG using immunoassay. Positive serum pregnancy test is defined as serum β-hCG concentration >10 mU/mL. The estimated period of time is 3 menstrual cycles (total of 9-15 weeks) or till pregnancy occurs whichever came first.
Change of Clinical pregnancy rate | The estimated period of time is 3 menstrual cycles with each menstrual cycle ranging from 3-5 weeks in duration (a total of 9-15 weeks) or till pregnancy occurs whichever came first.
  Patients with positive serum pregnancy test, defined as serum β-hCG concentration >10 mU/ml, were examined by abdominal ultrasonography, 6 weeks after the first day of their last menstrual period (LMP), using 3.5 MHz sector transducer (Esaote Mylab 50 Xvision Ultrasound, Italy) to detect an intrauterine gestational sac (Clinical pregnancy). Patients who failed to get pregnant were requested for follow up for 2 more consecutive cycles with the same protocol.
  The estimated period of time is 3 menstrual cycles (total of 9-15 weeks) or till pregnancy occurs whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mohamed Magdi Ammar, M.D., Principal Investigator — Saudi German Hospital - Madinah
Locations (1):
- Saudi German Hospital, Al Madīnah, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No